CLINICAL TRIAL: NCT07259473
Title: Factors Influencing Immunotherapy Response in Mismatch Repair Deficiency (dMMR) / Microsatellite Instability-High (MSI-H) Gastric/Gastroesophageal Junction Adenocarcinoma
Brief Title: Factors Influencing Immunotherapy Response in dMMR/MSI-H Gastric/Gastroesophageal Junction Adenocarcinoma
Acronym: Pre-CATALIS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xuefei.Wang, Chief of Department of Gastrointestinal Surgery, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-541R
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Gastric / Gastroesophageal Junction Adenocarcinoma; Mismatch Repair Deficient or MSI-High Solid Tumors; Immunotherapy
MeSH Terms: conditions — Turcot syndrome | interventions — Immunotherapy; Induction Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dMMR/MSI-H GC (Experimental): Immunotherapy with induction chemotherapy
  Interventions: Drug: Immunotherapy; Drug: Induction chemotherapy; Procedure: D2 radical gastrectomy

INTERVENTIONS:
Drug: Immunotherapy — Drug: Immune checkpoint inhibitors (ICIs), specifically PD-1 antibodies, PD-L1 antibodies, PD-1/CTLA-4 bispecific antibodies, or PD-1/CTLA-4 combination therapy.
  Regimen: 4 treatment cycles.
Drug: Induction chemotherapy — Drug: Oxaliplatin Regimen: 1 cycle Dosage: 130mg/m^2
Procedure: D2 radical gastrectomy — Curative-intent D2 radical gastrectomy is scheduled 4-6 weeks after completion of the fourth cycle.

SUMMARY:
dMMR/MSI-H is a key molecular subtype of gastric cancer, found in 8-22% of cases. It is typically associated with older age, female sex, distal tumor location, and intestinal histology (Lauren classification). While this subtype predicts better survival in locally advanced disease, its prognostic role in metastatic settings is less clear.

Notably, dMMR/MSI-H tumors are often resistant to conventional chemotherapy. Conversely, they demonstrate exceptional sensitivity to immunotherapy. This has led to effective strategies using immune checkpoint inhibitors, either alone or combined with chemotherapy, in both neoadjuvant and advanced disease settings.

However, key challenges remain. Prospective data are largely from Western populations, leaving the efficacy in Asian patients-who bear a high disease burden-less defined. Furthermore, about half of dMMR/MSI-H patients exhibit primary or acquired resistance to immunotherapy. A deeper understanding of the tumor-immune dynamics during treatment is crucial to uncover resistance mechanisms and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 85 years.
* Histologically confirmed gastric cancer or adenocarcinoma of the esophagogastric junction (only Siewert types II and III are included).
* dMMR status confirmed by immunohistochemistry (IHC) or MSI-H status confirmed by PCR/NGS.
* Tumor clinical staging meeting the following criteria:

cT≥2, any N, M0, assessed by the investigator as potentially resectable and planned for preoperative treatment followed by surgery.

* Willing to receive treatment with immune checkpoint inhibitors (including, but not limited to, various PD-1 inhibitors, PD-L1 inhibitors, CTLA-4 inhibitors, PD-1/CTLA-4 bispecific antibodies, etc.), which may be combined with or without standard chemotherapy regimens for gastric cancer.

Exclusion Criteria:

* Tumor histology other than adenocarcinoma, such as squamous cell carcinoma, neuroendocrine carcinoma, etc.
* Presence of central nervous system metastases and/or leptomeningeal carcinomatosis.
* Prior antitumor therapy directed at the current gastric cancer (excluding palliative gastrointestinal bypass surgery performed to relieve obstructive symptoms).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete response | From the initiation of treatment to the date of surgery, an average of 14 weeks.
  The proportion of subjects exhibiting no residual tumor cells in the surgical specimen and the absence of positive lymph nodes (i.e., a pathological stage of ypT0N0).

SECONDARY OUTCOMES:
Major Pathological Response Rate | From the initiation of treatment to the date of surgery, an average of 14 weeks.
  The proportion of subjects with residual viable tumor cells accounting for <10% of the surgical specimen from the primary tumor site.
ypN stage | From the initiation of treatment to the date of surgery, an average of 14 weeks.
  Lymph-node status after neoadjuvant therapy (ypN stage) will be assessed according to the American Joint Committee on Cancer (AJCC) 8th edition staging system.
R0 resection rate | From the initiation of treatment to the date of surgery, an average of 14 weeks.
  The proportion of patients who undergo surgery with microscopically negative resection margins.
Event-free Survival | The time from the initiation of treatment until disease progression, disease recurrence, death from any cause, or 3 years since enrollment.
  The time from the subject's enrollment until disease progression, disease recurrence, or death from any cause.
Overall Survival | From the initiation of treatment until death from any cause or 3 years since enrollment.
  The time from the subject's enrollment until death from any cause.

IPD SHARING:
Plan to Share IPD: No
Informed consent forms did not include provisions for public data sharing